CLINICAL TRIAL: NCT06568016
Title: Multilevel Intervention to Improve Follow-up Colonoscopy Rates After Abnormal FIT Results in Large FQHC
Brief Title: A Clinic-wide Intervention (Primary Care-GI Connect) for Improving Rates of Colonoscopy After Abnormal Fecal Immunochemical Test Result in Patients at Federally Qualified Health Centers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-000532; NCI-2024-05892 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-000532 (Other: UCLA / Jonsson Comprehensive Cancer Center); P30CA016042 (NIH)
Record Dates: First submitted 2024-07-29; First posted 2024-08-23 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods; Interviews as Topic; Patient Navigation; Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (usual care) (Active Comparator): Patients receive clinical care consistent with current practice at NEVHC. Patients have their EHRs reviewed monthly by the Primary Care FIT Tracker for abnormal FIT results and patients with abnormal FIT results receive standardized communication from FIT QI champions about their results and receive a referral to gastroenterology.
  Interventions: Other: Best Practice; Other: Communication Intervention; Other: Electronic Health Record Review; Other: Interview; Other: Referral
- Arm II (Usual care + Primary Care - GI Connect) (Experimental): Patients receive clinical care consistent with current practice at NEVHC as described in Arm I. Patients also receive enhanced GI care coordination from GI liaisons, who generate GI FIT Tracker reports and use the GI FIT Tracker reports to follow patients with abnormal FIT results. Patients receive navigation services including contact from GI liaisons about making a GI appointment and enhanced communication between GI specialists and the NEVHC. Patients receive referral to gastroenterology following a standardized referral template and receive colonoscopy education including an informational sheet at the time of referral and a 20-minute pre-colonoscopy educational video. Patients receive a text message at the time of colonoscopy referral emphasizing the importance of colonoscopy after abnormal FIT result.
  Interventions: Other: Best Practice; Other: Communication Intervention; Other: Coordination; Other: Educational Intervention; Other: Electronic Health Record Review; Other: Informational Intervention; Other: Interview; Behavioral: Patient Navigation; Other: Referral; Other: Text Message-Based Navigation Intervention

INTERVENTIONS:
Other: Best Practice — Receive clinical care consistent with current practice
  Other Names: standard of care; standard therapy
Other: Communication Intervention — Receive standardized communication from FIT QI champion
Other: Communication Intervention — Receive coordination from GI liaisons
  Arms: Arm II (Usual care + Primary Care - GI Connect)
Other: Coordination — Receive enhanced GI care coordination
  Arms: Arm II (Usual care + Primary Care - GI Connect)
Other: Educational Intervention — Watch pre-colonoscopy educational video
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm II (Usual care + Primary Care - GI Connect)
Other: Electronic Health Record Review — Undergo FIT result review by Primary Care FIT Tracker
Other: Electronic Health Record Review — Ancillary studies
Other: Informational Intervention — Undergo generation and review of GI FIT Tracker report
  Arms: Arm II (Usual care + Primary Care - GI Connect)
Other: Informational Intervention — Receive informational sheet
  Arms: Arm II (Usual care + Primary Care - GI Connect)
Other: Interview — Ancillary studies
Behavioral: Patient Navigation — Receive navigation from GI liaisons
  Other Names: Patient Navigator Program
  Arms: Arm II (Usual care + Primary Care - GI Connect)
Other: Referral — Receive referral
  Other Names: Referred
  Arms: Arm I (usual care)
Other: Referral — Receive referral per standardized template
  Other Names: Referred
  Arms: Arm II (Usual care + Primary Care - GI Connect)
Other: Text Message-Based Navigation Intervention — Receive follow-up text message
  Other Names: Automated Text Message-Based Navigation; Text Message-Based Navigation
  Arms: Arm II (Usual care + Primary Care - GI Connect)

SUMMARY:
This clinical trial evaluates a clinic-wide intervention called Primary Care-Gastrointestinal (GI) Connect for improving follow-up colonoscopy rates in patients at a Federally Qualified Health Center (FQHC) who have an abnormal fecal immunochemical test (FIT) result. Colorectal cancer screening reduces colorectal cancer incidence and mortality but is underutilized.The most accessible, feasible, and common colorectal cancer screening modality for average-risk individuals in low resource settings such as FQHCs is the stool-based FIT. However, the benefit of FIT screening on colorectal cancer risk is realized only if individuals with abnormal FIT results undergo timely follow-up colonoscopy. Follow-up colonoscopy rates are low and there are many barriers to follow-up colonoscopy in safety net settings such as FQHCs. Effective interventions that are multi-component and improve care coordination are needed to improve abnormal FIT follow-up rates in FQHCs. The Primary Care-GI Connect intervention includes components that enhance care coordination, standardize the referral process, and engage both primary care and specialist physicians. This clinic-wide intervention may improve rates of follow-up colonoscopy after abnormal FIT results in patients seen at FQHCs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Conduct a pragmatic, cluster randomized trial in 6 clinics (1500 patients) within a multi-site FQHC system to compare the effectiveness of the multilevel FQHC-GI care coordination intervention ("Primary Care-GI Connect "; 3 clinics, 750 patients) to the usual care condition (3 clinics, 750 patients) on receipt of a colonoscopy within 6 months of an abnormal FIT.

II. Systematically assess the quality of intervention implementation to understand the feasibility and relative importance of intervention elements as guided by the Multilevel Health Outcomes Framework.

III. Measure the incremental cost-effectiveness of the Primary Care-GI Connect intervention compared to usual care to understand the potential value, feasibility, and potential for dissemination.

OUTLINE: Northeast Valley Health Corporation (NEVHC) clinics are randomized to 1 of 2 arms.

ARM I: Patients receive clinical care consistent with current practice at NEVHC. Patients have their electronic health records (EHRs) reviewed monthly by the Primary Care FIT Tracker for abnormal FIT results and patients with abnormal FIT results receive standardized communication from FIT quality improvement (QI) champions about their results and receive a referral to gastroenterology.

ARM II: Patients receive clinical care consistent with current practice at NEVHC as described in Arm I. Patients also receive enhanced GI care coordination from GI liaisons, who generate GI FIT Tracker reports and use the GI FIT Tracker reports to follow patients with abnormal FIT results. Patients receive navigation services including contact from GI liaisons about making a GI appointment and enhanced communication between GI specialists and the NEVHC. Patients receive referral to gastroenterology following a standardized referral template and receive colonoscopy education including an informational sheet at the time of referral and a 20-minute pre-colonoscopy educational video. Patients receive a text message at the time of colonoscopy referral emphasizing the importance of colonoscopy after abnormal FIT result.

ELIGIBILITY:
Inclusion Criteria:

* 6 adult care NEVHC clinic sites

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Follow-up colonoscopy rates | At 6 months
  Evaluated in patients with an abnormal fecal immunochemical test (FIT) result using electronic health record data. Will use a difference-in-differences approach, assessing whether change in completion rates from baseline to the implementation period differs between the intervention and usual care conditions, thus accounting for potential differences among clinics pre-implementation. Will fit a mixed effects logistic regression model with a dependent variable of patient-level colonoscopy completion within 6 months (yes/no).
Implementation quality: fit tracker | Monthly intervals up to 3 years
  The Investigators will measure the percent of cases for which the FIT tracker is used, as well as its use for each step in the process. For these measures, we will also measure time to completion.
Implementation quality: patient notification | Monthly intervals up to 3 years
  The Investigators will measure both the percent of patients who are notified of their abnormal results as well as the time to notification.
Implementation quality: patient referral | Monthly intervals up to 3 years
  The Investigators will measure the percent of patients who receive a referral.
Implementation quality: Time to patient referral | Monthly intervals up to 3 years
  The Investigators will measure the time to patient referral.
Implementation quality: use of referral template as percent completion of interventions | Monthly intervals up to 3 years
  The Investigators will measure the percent completion of interventions for patients at each step.
Implementation quality: referral template in time to completion | Monthly intervals up to 3 years
  The Investigators will measure the time to completion of interventions.
Implementation quality: patient education | Monthly intervals up to 3 years
  The Investigators will measure the percent of cases in which patient education is delivered.
Implementation quality: patient education | Monthly intervals up to 3 years
  The Investigators will measure the time to delivery of patient education when it is offered.
Implementation quality: Patient attendance: completion of a pre-colonoscopy visit | Monthly intervals up to 3 years
  The Investigators will measure the percent of patients who complete a pre-colonoscopy visit.
Implementation quality: time to completion of a pre-colonoscopy visit | Monthly intervals up to 3 years
  The Investigators will measure the time to completion of a pre-colonoscopy visit.
Implementation quality: receipt of colonoscopy and pathology results at Northeast Valley Health Corporation | Monthly intervals up to 3 years
  The Investigators will measure the percent of patients for which colonoscopy and pathology results are received at NEVHC.
Implementation quality: receipt of colonoscopy and pathology results at Northeast Valley Health Corporation over time | Monthly intervals up to 3 years
  The Investigators will measure the time to retrieval of colonoscopy and pathology results received at NEVHC.
Cost-effectiveness | Up to 3 years
  Will use standard cost-effectiveness techniques (including time discounting) to conduct an incremental cost-effectiveness analysis, measuring the Incremental Cost-Effectiveness Ratio of the usual care and Primary-care GI connect intervention conditions.

SECONDARY OUTCOMES:
Time to colonoscopy | 0-24 months
  The Investigators will use a difference-in-differences approach, assessing whether change in completion rates from baseline to the implementation period differs between the intervention and usual care conditions, thus accounting for potential differences among clinics pre-implementation. Will fit a mixed effects logistic regression model with a dependent variable of patient-level colonoscopy completion.
Follow-up colonoscopy rates | At 9 months and at 12 months
  Evaluated in patients with an abnormal FIT result using electronic health record data. Will use a difference-in-differences approach, assessing whether change in completion rates from baseline to the implementation period differs between the intervention and usual care conditions, thus accounting for potential differences among clinics pre-implementation. Will fit a mixed effects logistic regression model with a dependent variable of patient-level colonoscopy completion within 9 months (yes/no).
Factors associated with Implementation | At pre-intervention (1-2 years) and at the implementation midpoint (3-4 years)
  The Investigators will use the Organizational Readiness to Implement Change tool to measure responses from clinic stakeholders at each site. This is a standardized tool.
Reported challenges to implementation | Up to 3 years
  In qualitative interviews with stakeholders and on standardized forms, we will learn about major challenges to implementation across clinics and over time. These will be qualitative data.
Intervention adaptations | Up to 3 years
  In qualitative interviews with stakeholders, we will learn whether there were any changes we need to be intended intervention components.
Clinic and provider factors | At pre-intervention (1-2 years) and at the implementation midpoint (3-4 years)
  The Investigators will use EHR data to measure clinic size, location, staffing, resources, number of providers, number of patients to evaluate associations with successful intervention implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Folasade P May, MD, PhD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University of California at Los Angeles, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California